CLINICAL TRIAL: NCT05739799
Title: Compariosn of Effectiveness of Diode Laser System Versus Intense Pulse Light (IPL) in The Treatment of Unwanted Hair
Brief Title: To Comapre The Effectiveness of Two Lasers in The Treamment of Unwanted Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Sara Ilyas, Principal Investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMH-ETH-18-DERM-22
Record Dates: First submitted 2023-01-18; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hirsuitism
MeSH Terms: conditions — Hirsutism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Intense pulse light laser (Active Comparator): IPL laser Patients in Group A received intense pulse light (IPL) frequency of 690. A total of three sessions were carried out one month apart, and hair reduction was assessed by seeing thickness of hair and by counting the number of hair follicles in a 1cm2 area on each side of the face before the first session and at the 4th month. A consultant dermatologist assessed the reduction in hair count on the affected side of face at the end of last session. Patients' response and any adverse effects experienced by patients' were recorded
  Interventions: Procedure: IPL
- Group B Diode laser (Active Comparator): Diode laser patients in Group B received diode laser treatment system. Diode laser was employed using triple wavelength (1064, 810 and 755 mm). A total of three sessions were carried out one month apart, and hair reduction was assessed by seeing thickness of hair and by counting the number of hair follicles in a 1cm2 area on each side of the face before the first session and at the 4th month. A consultant dermatologist assessed the reduction in hair count on the affected side of face at the end of last session. Patients' response and any adverse effects experienced by the patients were recorded.
  Interventions: Procedure: Diode

INTERVENTIONS:
Procedure: IPL — Patients in Group A received intense pulse light (IPL) frequency of 690. A total of three sessions were carried out one month apart, and hair reduction was assessed by seeing thickness of hair and by counting the number of hair follicles in a 1cm2 area on each side of the face before the first session and at the 4th month. A consultant dermatologist assessed the reduction in hair count on the affected side of face at the end of last session. Patients' response and any adverse effects experienced by patients' were recorded.
  Arms: Group A Intense pulse light laser
Procedure: Diode — patients in Group B received diode laser treatment system. Diode laser was employed using triple wavelength (1064, 810 and 755 mm). A total of three sessions were carried out one month apart, and hair reduction was assessed by seeing thickness of hair and by counting the number of hair follicles in a 1cm2 area on each side of the face before the first session and at the 4th month. A consultant dermatologist assessed the reduction in hair count on the affected side of face at the end of last session. Patients' response and any adverse effects experienced by the patients were recorded.
  Arms: Group B Diode laser

SUMMARY:
A total of 60 female patients (30 patients in each group) with unwanted facial hair diagnosed by a consultant dermatologist were included in this study. In Group A patients were subjected to intense pulse light therapy while patients in Group B were subjected to diode laser for three sessions one month apart. Effectiveness in both groups was ascertained in terms of hair reduction, less adverse effects, side effects and patients' satisfactory response at the end of final session.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with hirsuitism were included in the study.

Exclusion Criteria:

* tendency to develop hypertrophic scarring/keloid,
* underwent any treatment for unwanted facial hair in last two years
* pregnant/lactating women
* with hormonal imbalance and PCOS were also not in included in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of diode and IPL laser in hirsuitism | 12 weeks
  A total of 60 female patients (30 patients in each group) with unwanted facial hair diagnosed by a consultant dermatologist were included in this study. In Group A patients were subjected to intense pulse light therapy while patients in Group B were subjected to diode laser for three sessions one month apart. Effectiveness in both groups was ascertained in terms of hair reduction, less adverse effects, side effects, and patients' satisfactory response at the end of final session.After the "response at the end of final session the total duration of the therapy will be 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Ilyas, Abbottābād, Kpk, Pakistan